CLINICAL TRIAL: NCT03581682
Title: Tele-Clinic Visits in Pediatric Marfan Patients Using Parental Echo: The Future?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Seda Tierney, Associate Professor of Pediatrics, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 42159
Record Dates: First submitted 2018-06-18; First posted 2018-07-10 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Marfan Syndrome
MeSH Terms: conditions — Marfan Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele-Visit Using Parental Home Echo (Experimental): All parents will have hands-on echo training. We will test if a tele-visit using parental home echo is clinically reliable compared to an on-site clinic visit, costs less, and improves parental sense of empowerment.
  Interventions: Other: Tele-Clinic Visits Using Parent-Acquired Echos

INTERVENTIONS:
Other: Tele-Clinic Visits Using Parent-Acquired Echos — Every patient will have a tele-visit and an on-site clinic visit 1 day apart 3-6 months after the training session. Parents will have a 1-hour hands-on training session to acquire basic echo images on their children with the same hand-held device that they will use during the tele-visit. The parents will also have an in-service on how to take weight, height, and blood pressure measurements, and how to use the digital stethoscope.
  A tele-visit will be schedule a day prior to the patient's regularly scheduled clinic visit. Tele-visit elements will include interim medical history by the parent and patient, and weight, height, vital signs, digital cardiac auscultation, and home echo, all obtained by the parent. Two MFS physicians, following our routine MFS care protocol, will administer either the tele-visit or on-site clinic visit, masked to the findings of the other.

SUMMARY:
Marfan syndrome (MFS), a connective tissue disorder seen in 1 in 3,000 individuals, causes progressive aortic root dilation that can result in aortic dissection and sudden death. Clinical care focuses on monitoring the aortic root by serial echocardiography (echo) to guide medical treatment and elective aortic root surgery in a specialized clinic every 6-12 months. This monitoring protocol, coupled with surgical intervention, has doubled the median life expectancy which was previously only 32 years. However, this surveillance carries significant health care costs at >$50 million dollars/year on echos alone (at $3-4K each) in children and adolescents in the US, as well as substantial burden on families residing far from specialized centers. A clinic visit delivered to MFS patients via live-video conferencing at home (tele-visit) could shift this paradigm, if a home echo could be obtained.

Here, the investigator will train parents of Pediatric Marfan patients to take echo images using a hand held device, height, weight, blood pressure, medical history, and listen to the heart of their child. Then, the investigators will ask them to take the equipment home and collect the same data at home during a tele-clinic visit, with further instruction by the study team through secure live-video conferencing.

DETAILED DESCRIPTION:
In the proposed intervention, every patient (n=60) will have a tele-visit and an on-site clinic visit 1 day apart. Parents will have a 1-hour hands-on training session to acquire basic echo images on their children with the same hand-held device that will be used during the tele-visit. Tele-visit elements will include interim medical history by the parent and patient, and weight, height, vital signs, digital cardiac auscultation, and home echo (transferred via Internet for remote interpretation), all obtained by the parent. Two MFS physicians, following our routine MFS care protocol, will administer either the tele-visit or on-site clinic visit, masked to the findings of the other. Two independent echo readers will analyze home and clinic echos to measure reproducibility.

ELIGIBILITY:
Inclusion Criteria:

* 5-19 years of age (patient)
* seen in at least 2 prior clinic visits
* Marfan syndrome by revised Ghent criteria
* presence of parent at home

Exclusion Criteria:

* prior aortic surgery
* known cardiomyopathy
* known arrhythmia
* aortic root > 4.5 cm in prior clinic visit
* pregnancy

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Percent of tele-visits with a clinical visit match-score of ≥13/15 points | 3-6 months
  This scoring system was determined after surveying pediatric MFS physicians nationwide and includes these sections: Echo, vital signs, height and weight, interim medical history, cardiac auscultation, and determination of follow up time and medication dose/type.

SECONDARY OUTCOMES:
To test if a tele-visit using parental home echo costs less than an on-site clinic visit. | 3-6 months
  The outcome will be the costs of tele-visit and clinic visit. Two cost components will be estimated and combined costs will be compared: (1) Payer cost: Actual cost to deliver a tele-visit with home echo (as it is not currently covered by insurance) vs.
  Medical or private insurance reimbursement rates for clinic visit with an echo; and (2) Patient-cost: time and travel costs for parents.
To test if a tele-visit using parental home echo costs less than an on-site clinic visit. | 3-6 months
  Secondary outcome will be lost school time for the patient.
To determine if this intervention increases parental sense of empowerment. | 3-6 months
  The outcome will be the change in Family Empowerment Score (a validated questionnaire to assess empowerment in parents of children with illness) from study start to study end.
To determine if this intervention increases parental sense of empowerment. | 3-6 months
  Secondary outcomes will be parent/patient satisfaction survey results for televisits and clinic visits using the CAHPS survey for Children, as well as patient, parent and physician interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Tierney, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen A, Punn R, Collins RT, Chen JH, Stauffer KJ, Wang R, Alexander S, MacMillen Lechich K, Murphy DJ, Chung S, Selamet Tierney ES. Tele-Clinic Visits in Pediatric Patients with Marfan Syndrome Using Parentally Acquired Echocardiography. J Pediatr. 2021 May;232:140-146. doi: 10.1016/j.jpeds.2021.01.004. Epub 2021 Jan 13. PMID 33453199